CLINICAL TRIAL: NCT03189290
Title: Study of the QUadratus Lumborum Bloc in Total Hip ARthroplasty: Efficacy and Safety
Acronym: SQUARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9798
Record Dates: First submitted 2017-05-05; First posted 2017-06-16 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain; Total Hip Replacement
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ropivacaine (Active Comparator): Active Comparator: ropivacaine group
  - Before general anaesthesia, ultrasound guided Quadratus Lumborum Block (QLB) will be performed with 30 mL 0.33% Ropivacaine
  Interventions: Procedure: posterior Quadratus Lumborum Block (QLB)
- placebo (Placebo Comparator): Sham Comparator: saline group
  - Before general anaesthesia, ultrasound guided Sham Quadratus Lumborum Block (QLB) will be performed with 30 mL saline.
  Interventions: Procedure: posterior Quadratus Lumborum Block (QLB)

INTERVENTIONS:
Procedure: posterior Quadratus Lumborum Block (QLB) — Procedure (experimental): ultrasound guided posterior Quadratus Lumborum Block (QLB) Procedure (experimental): Sham Block

SUMMARY:
The purpose of this prospective research study is to determine the best way to manage post-operative pain after a total hip arthroplasty. Currently, there is no standard of care for managing post-operative pain in these patients. The quadratus lumborum block (QLB) first described by Blanco in 2007, is a promising technique in this indication: recently, there is a growing evidence for the use of the QLB as an alternative technique for pain management after hip surgery.

DETAILED DESCRIPTION:
A sample size of 100 patients (50 per group) was calculated based on 20% reduction in morphine consumption with 0.05% significance and a power of 0.8.

After ethical committee approval, eligible patients scheduled to have a fast-track total hip arthroplasty are screened during preoperative evaluation clinic. Informed written consent will be obtained from all patients during pre-anesthesia visit the day before surgery (J-1). Consenting patients will be randomized the day of surgery (J0) to undergo QLB with ropivacaine ("ropivacaine group") or normal saline ("saline group").

Before general anesthesia, all patients will have a needle-insertion posterior to the quadratus lumborum muscle avec injection of either ropivacaine in the "ropivacaine group" or normal saline in the "saline group".

After general anesthesia induction, dexamethasone and ketamine will be given to all patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Classification Status (ASA) I to III
* Age ≥ 18 years
* Scheduled for fast-track total hip arthroplasty
* Written informed consent
* Patient covered by health insurance Exclusion Criteria
* Protected patients or patients incapable of giving written informed consent
* Pregnant or breastfeeding woman
* Vulnerable adult
* Contraindication for fast-track surgery
* Inability to comprehend or participate in pain scoring scales
* Allergy to study drugs
* Severe coagulopathy
* Chronic kidney disease with glomerular filtration rate (GFR) ≤ 30 mL/min (estimated by the Cockcroft & Gault formula)
* Chronic pain (treated by nonsteroidal anti-inflammatory drugs, opioids, neuroleptic drugs, antidepressant or anticonvulsants)
* Peripheral neuropathy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of the posterior quadratus lumborum block (QLB) versus placebo on morphine consumption during the first 24 hours after a total hip arthroplasty | the first 24 hours after a total hip arthroplasty

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIBOULET, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Lapeyronie Teaching Hospital Montpellier, Montpellier, Occitanie, France